CLINICAL TRIAL: NCT03493217
Title: A Multicenter, Open-label Study to Evaluate the Safety and Efficacy of ICP-022 in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL) / Small Lymphocytic Lymphoma (SLL)
Brief Title: A Study to Evaluate ICP-022 in Patients With CLL/ SLL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00103
Record Dates: First submitted 2018-03-19; First posted 2018-04-10 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: CLL/SLL

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-022 (Experimental): Two regimens of ICP-022 (High and low dose QD) are designed for study Part I to determine RP2D. The RP2D determined will be used in Part II to further evaluate the preliminary efficacy of ICP-022 in Chinese subjects with R/R CLL/SLL.
  Interventions: Drug: ICP-022

INTERVENTIONS:
Drug: ICP-022 — The drug product is a white, round, uncoated tablet.

SUMMARY:
The phase I/II clinical study is to investigate the safety, tolerability and efficacy of ICP-022 in R/R CLL/SLL patients.

DETAILED DESCRIPTION:
Part I: Safety evaluation -2 regimens of ICP-022 (High and low dose QD) are designed for safety assessment. The recommended dose of phase II clinical study will be determined according to the Part I results.

Part II: Dose expansion -Anti-tumor effects of ICP-022 in Chinese patients with R/R CLL/SLL will be evaluated in approximately 80 subjects. The recommended Phase 2 dose will be used in the Part II.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with the age more than 18 years
* Subjects with confirmed diagnosis of CLL/SLL following IWCLL2008 criteria
* Refractory or relapsed CLL/SLL who have received at least one prior therapy
* At least two measurable tumors of greater than 1.5 centimeter in long axis by contrast-enhanced CT/MRI
* ECOG performance status of 0-2
* Documented failure to achieve at least partial response (PR) or documented disease progression after response to, the most recent treatment regimen.There are medicalrecords confirming that the disease has not responded to the mostrecent treatment (complete and partial remission) or that thedisease has progressed after remission
* Subjects who meet the following laboratory parameters:

  * Absolute neutrophil count (ANC) ≥ 0.75×109/L, Platelet count ≥ 50×109/L independent of growth factor support within 7 days of the first dose of study drug
  * Total bilirubin ≤ 2× ULN (unless due to Gilbert's syndrome); AST or ALT ≤ 2.5 ULN; Creatinine ≤ 1.5 ULN; Amylase ≤ 1.5 ULN
  * International normalized ratio (INR) ≤ 1.5 ULN and activated partial thromboplastin time (APTT) ≤ 1.5 ULN
* Life expectancy ≥ 4 months
* Able to provide signed written informed consent

Exclusion Criteria:

* History of other active malignancies within 5 years of study entry, unless cured without evidence of relapse or metastasis
* Current or history of lymphoma involved central nervous system
* Any history of Richter's transformation
* Prior corticosteroids (at dosages equivalent to prednisone > 20 mg/day) given with anti-neoplastic intent within 7 days, prior chemotherapy, targeted therapy, radiation therapy, or antibody based therapies or anti-cancer TCM within 4 weeks of the start of study drug.
* Non-hematological toxicity must be recovered to ≤ Grade 1 from prior anti-cancer therapy (except alopecia)
* Current Clinically significant cardiovascular disease including:

  * Any class 3 or 4 cardiac disease such as arrhythmia, congestive heart failure or myocardial infarction defined by the New York Heart Association Functional Classification, or left ventricular ejection fraction (LVEF) < 50%
  * Primary cardiomyopathy
  * Clinical significant QTc prolong history or QTc>470ms (female) QTc>450ms (male)
  * Uncontrolled hypertension
* Subjects with active bleeding within 2 months of study start or currently taking anticoagulant/antiplatelet drugs
* Urine protein ≥ 2+ and quantitation ≥ 2g/24hours
* History of deep vein thrombosis or pulmonary embolism
* Disease significantly affecting gastrointestinal function such as dysphagia, chronic diarrhea, intestinal obstruction, or resection of the stomach
* Prior allogeneic stem cell transplant within 6 months prior to first dose of study drug or related active infection
* Prior organ or allogeneic hematopoietic stem cell transplant within 6 months prior to first dose of study drug
* Major surgery within 6 weeks of screening, except for diagnostic test or vascular access setup
* Known active infection with HBV, HCV or HIV or any uncontrolled active systemic infection
* Any history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe lung function impairment
* Prior exposure to a BTK inhibitor or PI3K, SYK, bcl-2 inhibitors
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Any mental or cognitive disorder, unable to understand and comply with the requirements of the study
* Drug abuser or alcoholics
* Lactating or pregnant women, or women who will not agree to use contraception during the study and for 180 days after the last dose of study drug if sexually active and able to bear children
* Requires treatment with moderate or strong cytochrome P450 family 3, subfamily A (CYP3A) inhibitors or strong CYP3A inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
1.Objective response rate (ORR) | Up to 3 years
  The efficacy measured by overall response rate (ORR) in Part II. Efficacy was evaluated by researchers according to IWCLL2008standard and update standard (Hallek, 2012), which was defined as complete remission (CR) of CLLsubjects, complete remission with incomplete bone marrow recovery (CRi), or partial remission (PR),including nodular partial remission (nPR) and partial remission with lymphocytosis (pr-l).SLL subjectsachieved complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Occurrence of adverse events and serious adverse events according to NCI-CTCAE 4.03 grading criteria | Up to 3 years
  The safety and tolerability of ICP-022 measured by the occurrence of adverse events and serious adverse events according to NCI-CTCAE 4.03 grading criteria in Part I
TTR | Up to 3 years
  The efficacy measured by time to response (TTR) in Part II
TTP | Up to 3 years
  The efficacy measured by time to progression (TTP) in Part II
PFS | Up to 3 years
  The efficacy measured by progression free survival (PFS) in Part II
DOR | Up to 3 years
  The efficacy measured by duration of response (DOR) in Part II
OS | Up to 3 years
  The efficacy measured by overall survival (OS) in Part II

CONTACTS AND LOCATIONS:
Overall Officials: Jianyong Li, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (25):
- China (25):
  - Anhui Province Cancer Hospital, Hefei, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Henan Tumor Hospital, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The second affiliated hospital of dalian medical university, Dalian, Liaoning
  - Qilu Hosptial of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Xinhua hospital affiliated to medical college of Shanghai jiao tong university, Shanghai, Shanghai Municipality
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - The Chinese Academy of Medical Sciences Hematology Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Second affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No